CLINICAL TRIAL: NCT05365477
Title: Randomized Trial of Empiric Versus Selective Prevention Strategies for Kidney Stone Disease
Brief Title: Empiric Versus Selective Prevention Strategies for Kidney Stone Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, David Penson, Professor and Chair, Department of Urology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 200238
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Kidney Stones; Nephrolithiasis
Keywords: Prevention
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Empiric Therapy (Active Comparator): Diet intervention and drug intervention not based on 24 hour urine results
  Interventions: Behavioral: Empiric Therapy: Diet; Drug: Empiric Therapy: Drug
- Selective Therapy (Experimental): Diet intervention and drug intervention based on 24 hour urine results
  Interventions: Behavioral: Selective Therapy: Diet; Drug: Selective Therapy: Drug

INTERVENTIONS:
Behavioral: Empiric Therapy: Diet — Diet: High water intake - at least 2.5 liters daily Reduce sugar-sweetened cola intake to ≤3 cans per week. Reduce salt intake to <2000mg sodium daily Reduce red meat intake to two 4-ounce portions per week Normal calcium intake: 3 servings of dairy products (or their equivalents) per day Increase vegetable and fruit intake to ≥5 servings per day Reduce oxalate intake to <100 mg/day
  Arms: Empiric Therapy
Drug: Empiric Therapy: Drug — Drug(s): indapamide 1.25mg and potassium citrate 15mEq daily.
  Arms: Empiric Therapy
Behavioral: Selective Therapy: Diet — Diet:
  Volume <2.5L Increase fluid intake to ≥ 2.5L/d, based on specific urine volume
  Calcium >250mg male, >200mg female Reduce red meat intake to two 4-oz portions/wk; reduce sodium intake to<2000mg/d, avoid vitamin D + calcium supplements
  Oxalate >40mg Reduce dietary oxalate intake to <100 mg/d; increase fiber intake to 25-35 g/d
  Citrate <450mg male, <550mg female Reduce red meat intake to two 4-oz portions/wk; increase fruit and vegetable intake to ≥5 svgs/d
  pH<5.8 Reduce red meat intake to two 4-oz portions/wk; increase fruit and vegetable intake to ≥5 svgs/d
  Uric acid >800mg male, >750mg female Reduce red meat intake to two 4- oz portions/wk; increase fruit and vegetable intake to ≥5 svgs/d
  Sodium >150mmol Reduce sodium intake to <2000mg/d
  Sulfate > 80mEq or urine urea nitrogen >14g Reduce red meat intake to three 3-4 oz portions/wk; increase fruit and vegetable intake to ≥5 svgs/d
  Arms: Selective Therapy
Drug: Selective Therapy: Drug — Drug(s):
  For calcium >250mg male, >200mg female: indapamide 1.25mg and potassium chloride 20mEq. At 1 month if persistent, then increase to indapamide 2.5mg and potassium chloride 20mEq. For citrate <450mg male, <550mg female: potassium citrate 15mEq BID. At 1 month if persistent, then increase to potassium citrate 30mEq BID. For pH<5.8: potassium citrate 15mEq BID. At month if persistent, then increase to potassium citrate 30mEq BID. For uric acid >800mg male, >750mg female: allopurinol 300mg.
  If both elevated calcium and low pH: indapamide 1.25mg and potassium citrate 15mEq BID If both elevated calcium and low citrate: indapamide 1.25mg and potassium citrate 15mEq BID
  Arms: Selective Therapy

SUMMARY:
The aims of this study are to 1) Conduct a randomized clinical trial of selective versus empiric diet plus pharmacologic therapy in high-risk stone formers and 2) Determine adverse effects from, and adherence to selective and empiric strategies.

DETAILED DESCRIPTION:
Diet and pharmacologic interventions for preventing future kidney stone episodes are effective, however clinical guideline panels disagree on whether clinicians should perform selective therapy: performing 24-hour urine testing to guide choosing interventions to correct abnormal urinary parameters. The alternative strategy is empiric therapy: applying interventions without 24-hour urine testing. While 24-hour urine testing is considered the standard of care by nephrology and urology specialties for higher risk patients, the American College of Physicians does not recommend 24-hour urine testing.

This is a randomized clinical trial of selective versus empiric therapy for patients with presumed idiopathic calcium stone disease, representing >80% of the kidney stone population. The primary outcome is change in urinary supersaturation, which associates with symptomatic stone recurrence. We will recruit patients with presumed idiopathic calcium stone disease with at least 2 stone events within the previous 5 years. Participants will be randomly assigned to empiric diet plus thiazide with potassium citrate daily, or to selective diet plus pharmacologic therapy based on the 24-hour urine abnormalities identified at baseline and adjusted during follow-up. The primary outcomes will be the calculated calcium oxalate and calcium phosphate supersaturations. In addition, we will determine adverse effects from, and adherence to, selective and empiric strategies.

ELIGIBILITY:
Inclusion Criteria:

* Two or more symptomatic kidney stone events in the last 5 years
* Adult

Exclusion Criteria:

* Medullary sponge kidney or renal tubular acidosis
* Untreated urinary obstruction
* Primary hyperparathyroidism
* Primary hyperoxaluria
* Pregnancy
* Inflammatory bowel disease or bowel resection
* Sarcoidosis
* Cystinuria
* Prior stone composition with uric acid, struvite, cystine, carbonate apatite
* Use of specific medications (thiazides, topiramate, xanthine oxidase inhibitors, citrate, bicarbonate)
* Chronic kidney disease stage 3 or higher (eGFR<60)
* Gouty arthritis or 3 gout episodes in 1 year
* Known allergy to study medications
* Hypokalemia or hyponatremia at screening.
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-08-04 (Actual); Primary Completion 2025-10-17 (Actual); Study Completion 2025-10-17 (Actual)

PRIMARY OUTCOMES:
Calcium oxalate supersaturation | Baseline compared to two months
  Calculated calcium oxalate supersaturation in urine
Calcium phosphate supersaturation | Baseline compared to two months
  Calculated calcium phosphate supersaturation in urine

SECONDARY OUTCOMES:
Uric acid supersaturation | Baseline compared to two months
  Calculated uric acid supersaturation in urine
24hr urine parameters | Baseline compared to two months
  Urinary volume, calcium, oxalate, potassium, citrate, pH, uric acid, and sodium

OTHER OUTCOMES:
24hr urine parameters from baseline to month 1 | Baseline to 1 month
  Calculated urinary supersaturations of calcium oxalate, calcium phosphate, uric acid, and urinary volume, calcium, oxalate, potassium, citrate, pH, uric acid, and sodium
24hr urine parameters from month 1 to month 2 | 1 month to 2 months
  Calculated urinary supersaturations of calcium oxalate, calcium phosphate, uric acid, and urinary volume, calcium, oxalate, potassium, citrate, pH, uric acid, and sodium
Kidney stone events | Baseline to 2 months
  Assessment of short term kidney stone events by self report and clinical imaging, if available
Adverse events | Baseline to 2 months
  Assessment of adverse events - subjective and new hypokalemia, hyponatremia, hypomagnesemia, gouty arthritis or requiring uric acid lowering therapy, newly developed overt diabetes mellitus, allergic reactions, abnormal heart rate and blood pressure.
Diet adherence | Baseline to 2 months
  Food diaries
Medication adherence | Baseline to 2 months
  Pill counts

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Hsi, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-01-15): https://cdn.clinicaltrials.gov/large-docs/77/NCT05365477/ICF_000.pdf